CLINICAL TRIAL: NCT01535963
Title: A Pilot Study of Patient Satisfaction After Cutaneous Surgery
Brief Title: Patient Satisfaction in Cutaneous Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Other Study IDs: STU55818
Record Dates: First submitted 2012-02-07; First posted 2012-02-20 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cutaneous surgery: Patients undergoing cutaneous surgery

SUMMARY:
The primary objective of this study is to measure the overall level of satisfaction in patients after cutaneous surgery in 4 different categories, including the surgeon, facility, procedure and recovery and outcome.

DETAILED DESCRIPTION:
Secondary objectives are to identify factors associated with patient satisfaction level and determine the correlation between patient satisfaction and surgeon clinical perception.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Is in a self-reported stable health condition
* English speaking
* Is willing and has the ability to understand the study, provide informed consent and communicate with the investigator
* Recommended to have and scheduled for cutaneous surgery
* Agrees to follow-up at scheduled times

Exclusion Criteria:

* Unable to speak or read English
* Did not complete an 8th grade education
* A history of mental illness
* Any other disability or condition that would prevent completion of questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cutaneous surgery
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2012-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient rating | at time of visit
  Subjects will rate their satisfaction after cutaneous surgery in 4 different categories using 0-10 visual analog scales. The scale will be ~100 millimeters in length and each response will be given a value in millimeters. In addition, patients will answer an open-ended question about their level of satisfaction. Data will also be compared to previous data from patients after cutaneous surgery in the literature.

SECONDARY OUTCOMES:
Patient ranking | at time of visit
  Subjects will rank the factors determining satisfaction in order of importance using a ranking system for each aspect of care. In addition, the surgeon will rate their satisfaction level and give their perception on patient satisfaction and communication level using 0-10 visual analog scales

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States